CLINICAL TRIAL: NCT06506396
Title: Outcomes and Rehabilitation Needs of Patients With Hematologic Cancer Candidate for Hematopoietic Stem Cell Transplantation or CAR T-Cell Therapy: a Prospective Observational Study
Brief Title: Rehabilitation Needs for Hematologic Cancer Candidate for Hematopoietic Stem Cell Transplantation or CAR T-Cell Therapy
Acronym: HEMATOneeds
Status: Not yet recruiting | Type: Observational
Sponsor: University of Modena and Reggio Emilia (Other)
Collaborators: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Principal Investigator, Stefania Costi, Researcher, University of Modena and Reggio Emilia
Other Study IDs: 2024/0087161_26/06/2024
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Stem Cell Transplantation; Immunotherapy; CAR T-Cell Therapy
Keywords: Functional Status; Quality of life; Needs Assesment; Physical Conditioning, Human; Hematologic Neoplasms
MeSH Terms: conditions — Motor Activity; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with hematologic cancer scheduled to undergo HSCT or CAR T-cell therapy: The participants will be selected at the Hematology Unit of Azienda USL-IRCCS di Reggio Emilia, Northern Italy, two months prior to undergoing transplantation or CAR-T cell treatment. Eligible participants must meet the following inclusion criteria: have hematologic cancer and be scheduled for HSCT or CAR T-cell therapy; be at least 18 years old; able to provide informed consent and actively participate in the study; proficient in understanding and communicating in Italian.
  Patients who are unable to perform physical tests or have contraindications to movement will be excluded from the study

SUMMARY:
Hematopoietic Stem Cell Transplantation (HSCT) and CAR T-cell therapy are effective treatments for blood cancers, extending patients lives. However, these treatments can cause side effects like muscle weakness and fatigue. Recent findings suggest these issues can significantly affect patient quality of life during CAR T-cell therapy.

Patients undergoing HSCT and CAR T-cell therapy often face frequent infections and strong immune responses, requiring long periods of rest. This worsens their physical condition and impacts their quality of life, muscle strength, and fatigue levels. Minimizing these side effects is crucial to improve the well-being of patients undergoing these advanced treatments.

This study aims to assess the physical abilities (main goal) of patients preparing for HSCT or CAR T-cell therapy. It also aims to examine their quality of life and describe the symptoms and complications they may experience. The results will help identify rehabilitation needs for these patients.

DETAILED DESCRIPTION:
This is a prospective observational study following STROBE guidelines for observational studies in epidemiology. The study will take place at the Azienda USL-IRCCS di Reggio Emilia, Northern Italy.

Participants will include adults with blood cancer scheduled for HSCT or CAR T-cell therapy. They must be able to understand and speak Italian and make an informed decision to participate in the study.

Patients will be identified at the Hematology Unit of Azienda USL-IRCCS di Reggio Emilia. Medical records will be reviewed to confirm eligibility. Eligible patients will receive detailed information about the study and can decide to participate by signing a consent form.

The study will last 24 months, with an 8-month enrollment period and an 8-month follow-up. Approximately 20 participants will be enrolled based on the number of patients who received HSCT and CAR T-cell therapy in 2023.

Data on participants Sociodemographic and clinical characteristics will be collected at the start of the study. Complications and hospitalizations will be monitored after treatments to understand their impact on patients health.

This study aims to provide valuable insights into the rehabilitation needs of patients undergoing HSCT and CAR T-cell therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematologic cancer scheduled to undergo HSCT or CAR T-cell therapy;
* Age ≥18 years
* Able to provide informed consent to participate in the study
* Able to understand and participate in the study
* Able to understand and communicate in the Italian language

Exclusion Criteria:

• Patients who are unable to perform physical tests or have contraindications to movement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The potential participants will be selected at the Hematology Unit of the Azienda USL-IRCCS di Reggio Emilia among patients undergoing hematopoietic stem cell transplantation or CAR T-cell treatment, identified two months prior to their treatment.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Physical function | From enrollment up to 8 months later.
  Time up and go (TUG)
Phyical Function | From enrollment up to 8 months later.
  Short Physical Performance Battery (SPPB)

SECONDARY OUTCOMES:
Strength | From enrollment up to 8 months later.
  Handgrip strength test
Quality of life | From enrollment up to 8 months later.
  European Organization for Research and Treatment of Cancer QoL Questionnaire-C30 -QLQ C30. This questionnaire will be administered to assess participants' quality of life. It comprises one global scale, five functional scales, three symptom scales, and six single item scale.All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems
Fatigue | From enrollment up to 8 months later.
  Functional Assesment of Chronic IIlness Therapy-Fatigue.the total score range is 0 to 52. The general population mean score is 43. Lower scores indicate greater fatigue.
Activity of daily living | From enrollment up to 8 months later.
  Duke Activities Score Index (DASI).The DASI is a 12-item questionnaire that asses daily activities in the following domain: productivity, self-care, and leisure time. Total score ranges from 0 to 58.2. Higher scores indicate higher self-perceived functional ability.
Physical activity | From enrollment up to 8 months later.
  International Physical Activities Questionnarie_Short Form (IPAQ-SF).This self-reported questionnaire provides information on the intensity, duration, and frequency of various physical activities, offering valuable insights into participants' overall activity levels. In addition, Metabolic Equivalent of Tasks (METs) are used to classifies the level of patients' physical activity as low (<600 MET), moderate (from 600 to 3000 MET), or high (≥ 3000 MET)
KInesiophobia | From enrollment up to 8 months later.
  Tampa Scale of Kinesiophobia (TSK)The 17 item TSK total scores range from 17 to 68 where the lowest 17 means no or negligible kinesiophobia, and the higher scores indicate an increasing degree of kinesiophobia
Walking ability | From enrollment up to 8 months later.
  Functional Ambulation Category (FAC).Clinician-completed tick box of 5 broad categories of walking ability, ranges from independent walking outside (score 5) to non-functional walking (score 0).

OTHER OUTCOMES:
Compilcation | From Treatment up to 8 month
  Treatment complication
Legth of stay | From Treatment up to 8 month
  Days of hospitalisation

CONTACTS AND LOCATIONS:
Locations (1):
- AUSL-IRCCS di Reggio Emilia, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: No
IPD are sensible data and then will not be shared